CLINICAL TRIAL: NCT04397276
Title: A Phase 1 Study of JNJ-70218902, a T Cell Redirecting Agent, in Advanced Stage Solid Tumors
Brief Title: A Study of JNJ-70218902 in Participants With Advanced Stage Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108765; 70218902EDI1001 (Other: Janssen Research & Development, LLC); 2019-004885-16 (EudraCT Number); 2024-516351-40-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms
Keywords: metastatic Castration-Resistant Prostate Cancer (mCRPC); Prostate Cancer
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants with metastatic castration-resistant prostate cancer (mCRPC) will receive JNJ-70218902. The dose levels will be escalated sequentially based on the decisions of the Study Evaluation Team (SET) until the recommended Phase 2 Dose (RP2D) has been identified.
  Interventions: Drug: JNJ-70218902
- Part 2: Dose Expansion (Experimental): Participants with mCRPC will receive JNJ-70218902 at the RP2D determined in Part 1.
  Interventions: Drug: JNJ-70218902

INTERVENTIONS:
Drug: JNJ-70218902 — JNJ-70218902 will be administered.

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose(s) (RP2D[s]) and maximum tolerated dose (MTD) of JNJ-70218902 in Part 1, and to determine the safety of JNJ-70218902 RP2D(s) in Part 2.

DETAILED DESCRIPTION:
JNJ-70218902, the investigational drug, has been shown in pre-clinical studies to work by attaching to cancer cells and activating immune cells to kill these cancer cells. This study will be conducted in 2 parts: dose escalation (Part 1) and dose expansion (Part 2) and will enroll adult men with Metastatic Castration-Resistant Prostate Cancer (MCRPC). Study evaluations will include preliminary clinical efficacy, safety, pharmacokinetics, biomarkers and immunogenicity evaluations. This study is divided into 3 periods: screening, treatment and post-treatment. The total duration of the study will be 2.5 years approximately.

ELIGIBILITY:
Inclusion Criteria:

* Histology: Metastatic castration-resistant prostate cancer (mCRPC) with histologic confirmation of adenocarcinoma. Adenocarcinoma with small-cell or neuroendocrine features is allowed
* Measurable or evaluable disease
* Prior treatment with at least 1 prior novel androgen receptor (AR)-targeted therapy or chemotherapy
* If the participant is receiving treatment with gonadotropin-releasing hormone agonists or antagonist analogs (GnRH), this therapy must have been initiated prior to first dose of study drug and must be continued throughout the study
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Adequate organs functions

Exclusion Criteria:

* Known brain metastases
* Concurrent use of any other anticancer treatment or investigational agent for the treatment of advanced disease
* Toxicities related to prior anticancer treatments have not returned to Grade less than or equal to (<=) 1 or baseline, except for alopecia and vitiligo
* Solid organ or bone marrow transplantation
* Known allergies, hypersensitivity, or intolerance to JNJ-70218902 or its excipients
* Certain comorbidities

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 2.5 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part 1: Number of Participants with Dose-Limiting Toxicity (DLT) | Up to 21 days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Part 1 and Part 2: Number of Participants with AEs by Severity | Up to 2.5 years
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 with the exception of cytokine release syndrome (CRS), which will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of JNJ-70218902 | Up to 2.5 years
  Cmax is the maximum observed serum concentration of JNJ-70218902.
Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-70218902 | Up to 2.5 years
  Tmax is defined as time to reach maximum observed serum concentration.
Area Under the Serum Concentration-time Curve From t1 to t2 Time (AUC[t1-t2]) of JNJ-70218902 | Up to 2.5 years
  AUC(t1-t2) is defined as the area under the serum concentration-time curve from time t1 to t2.
Area Under the Concentration-time Curve From Time Zero to End of Dosing Interval (AUCtau) of JNJ-70218902 | Up to 2.5 years
  AUCtau is the measure of the serum drug concentration from time zero to end of dosing interval.
Minimum Observed Serum Concentration (Cmin) of JNJ-70218902 | Up to 2.5 years
  Cmin is the minimum observed serum concentration of JNJ-70218902.
Accumulation Ratio (RA) of JNJ-70218902 | Up to 2.5 years
  Accumulation Ratio (RA) is calculated as area under the plasma concentration-time curve from time zero to 24 hours (AUC [0-24]) value at steady state divided by AUC (0-24) value after first dose.
Systemic Cytokine Concentrations | Up to 2.5 years
  Cytokines concentration will be measured for biomarker assessment.
Serum Prostate Specific Antigen (PSA) Concentration | Up to 2.5 years
  Serum prostate specific antigen (PSA) concentration will be measured.
Number of Participants With Anti-JNJ-70218902 Antibodies | Up to 2.5 years
  Number of participants with anti-JNJ-70218902 antibodies will be assessed.
Objective Response Rate (ORR) | Up to 2.5 years
  ORR is defined as the percentage of participants who have a Partial Response (PR) or better according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 without evidence of bone progression according to Prostate Cancer Working Group 3 (PCWG3).
Duration of Response (DOR) | Up to 2.5 years
  Duration of response (DOR) will be calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the PCWG3 or RECIST version 1.1 response criteria, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- Canada (2):
  - BC Cancer Agency - Vancouver BC, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
- Israel (2):
  - Rambam Medical Center, Haifa
  - Sourasky Medical Center, Tel Aviv
- Spain (3):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency